CLINICAL TRIAL: NCT00778830
Title: An Asia Pacific Non-randomized, Open-label Phase II Study Evaluating the Safety and Efficacy of FOLFIRI Plus Cetuximab (Erbitux) or FOLFOX Plus Cetuximab as First-line Therapy in Subjects With KRAS Wild-type Metastatic Colorectal Cancer (APEC-Study)
Brief Title: Study Evaluating the Safety and Efficacy of FOLFIRI Plus Cetuximab or FOLFOX Plus Cetuximab as First-line Therapy in Subjects With KRAS Wild-type Metastatic Colorectal Cancer (APEC-Study)
Acronym: APEC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Pte. Ltd., Singapore (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62202-505
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Results first posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mCRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; IFL protocol; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetuximab plus FOLFIRI (Experimental)
  Interventions: Drug: Cetuximab; Drug: FOLFIRI
- Cetuximab plus FOLFOX (Experimental)
  Interventions: Drug: Cetuximab; Drug: FOLFOX

INTERVENTIONS:
Drug: Cetuximab — Cetuximab will be administered intravenously at a dose of 500 milligram per square meter (mg/m^2) biweekly on Day 1 of 14 days treatment cycle until disease progression, occurrence of unacceptable toxicity, or withdrawal of consent.
  Other Names: Erbitux
Drug: FOLFIRI — Irinotecan will be administered intravenously at a dose of 180 mg/m^2 along with folinic acid administration intravenously at a dose of 400 mg/m^2 (racemic) or 200 mg/m^2 (L-form) and 5-fluorouracil will be administered intravenously at a dose of 400 mg/m^2 bolus followed by a 46-hour continuous infusion of 2,400 mg/m^2 given biweekly until disease progression, death, or consent withdrawal.
  Arms: Cetuximab plus FOLFIRI
Drug: FOLFOX — Oxaliplatin will be administered intravenously at a dose of 100 mg/m^2 along with folinic acid administration intravenously at a dose of 400 mg/m^2 (racemic) or 200 mg/m^2 (L-form) and 5-fluorouracil administration intravenously at a dose of 400 mg/m^2 bolus followed by a 46-hour continuous infusion of 2,400 mg/m^2 given biweekly until disease progression, death, or consent withdrawal.
  Arms: Cetuximab plus FOLFOX

SUMMARY:
This is an open-label, non-randomized, multicenter Phase II study evaluating folinic acid + fluorouracil + irinotecan (FOLFIRI) plus cetuximab (Erbitux) or folinic acid + fluorouracil + oxaliplatin (FOLFOX) plus cetuximab as first-line therapy of patients with KRAS wild-type metastatic colorectal cancer.

Only subjects with k-ras oncogene (KRAS) wild-type tumors are eligible. Efficacy will be assessed every 8 weeks. Treatment will be continued until progressive disease or unacceptable adverse events occur. After the end of study treatment, information on further anticancer treatment and survival will be collected every 3 months.

ELIGIBILITY:
Inclusion Criteria:

Signed written informed consent

* Inpatient or outpatient subjects, 18 years of age
* Diagnosis of histologically confirmed adenocarcinoma of the colon or rectum
* Metastatic disease (M1)
* Life expectancy of at least 12 weeks
* Presence of at least 1 measurable index lesion (not lie in an irradiated area) by computed tomography (CT) scan or magnetic resonance imaging (MRI)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at study entry
* Effective contraception for both male and female subjects if the risk of conception exists
* White blood cell count greater than or equal to (>=) 3,000 per cubic millimeter (/mm^3) with neutrophils >=1,500/mm3, platelet count >=100,000/mm3, hemoglobin >=5.6 millimole per liter (mmol/L) (9 gram per deciliter [g/dL])
* Total bilirubin less than or equal to (<=) 1.5 x upper reference range
* Aspartate aminotransferase (AST) <=2.5 x upper reference range, or <=5 x upper reference range in case of liver metastasis
* Serum creatinine <=1.5 x upper reference range
* Recovery from relevant toxicity to previous treatment before study entry
* KRAS wild-type status of tumor tissue

Exclusion Criteria:

* Previous chemotherapy for colorectal cancer except adjuvant treatment if terminated >6 months before the start of treatment in this study
* Radiotherapy, surgery (excluding prior diagnostic biopsy) or any investigational drug in the 30 days before the start of treatment in this study
* Concurrent chronic systemic immune therapy, targeted therapy, anti-vascular endothelial growth factor (VEGF) therapy, or epidermal growth factor receptor (EGFR-) pathway targeting therapy not indicated in this study protocol
* Concurrent hormone therapy not indicated in this study protocol except for physiologic replacement or contraception
* Known hypersensitivity reaction to any of the components of study treatments
* Pregnancy (absence to be confirmed by beta human choriongonadotrophin [beta-hCG] test) or lactation period
* Brain metastasis and/or leptomeningeal disease (known or suspected)
* Clinically relevant coronary artery disease, history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease
* Peripheral neuropathy > grade 1
* Previous malignancy other than colorectal cancer in the last 5 years except basal cell cancer of the skin or preinvasive cancer of the cervix
* Known alcohol or drug abuse
* Medical or psychological conditions that would not permit the patient to complete the study or sign informed consent
* Participation in another clinical study within the past 30 days
* Significant disease which, in the investigator's opinion, would exclude the patient from the study
* Legal incapacity or limited legal capacity
* KRAS mutated status of tumor tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2009-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Pte. Ltd., Singapore
Locations (1):
- Research Site, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/Last subject (informed consent): February 2009/June 2012. Study completion date: April 2014. Clinical data cut-off: 31 March 2014. Subjects were recruited in 12 countries (Australia, China, Hong Kong, India, Indonesia, Korea, Malaysia, Singapore, Pakistan, Philippines, Taiwan and Thailand) across the globe in 43 centers.
Pre-assignment Details: Enrolled: 661 screened for eligibility; 372 were excluded (mainly non-fulfillment of inclusion or exclusion criteria). 289 subjects were assigned to the treatment groups.
Groups:
- Cetuximab Plus FOLFIRI: Cetuximab was administered intravenously at a dose of 500 milligram per square meter (mg/m^2) biweekly followed by Folfiri (Irinotecan administered intravenously at a dose of 180 mg/m^2 ,folinic acid administered intravenously at a dose of 400 mg/m^2 (racemic) or 200 mg/m^2 (L-form), 5-fluorouracil administered intravenously at a dose of 400 mg/m^2 bolus followed by a 46-hour continuous infusion at a dose of 2,400 mg/m^2) on Day 1 of 14 days treatment cycle until disease progression, occurrence of unacceptable toxicity, or withdrawal of consent.
- Cetuximab Plus FOLFOX: Cetuximab was administered intravenously at a dose of 500 milligram per square meter (mg/m^2) biweekly followed by Folfox (Oxaliplatin administered intravenously at a dose of 180 mg/m^2, folinic acid administered intravenously at a dose of 400 mg/m^2 (racemic) or 200 mg/m^2 (L-form), 5-fluorouracil administered intravenously at a dose of 400 mg/m^2 bolus followed by a 46-hour continuous infusion at a dose of 2,400 mg/m^2) on Day 1 of 14 days treatment cycle until disease progression, occurrence of unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | Cetuximab Plus FOLFIRI | Cetuximab Plus FOLFOX
Started | 101 | 188
Completed | 101 | 187
Not Completed | 0 | 1
Not completed — Ongoing at data cut-off | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population consisted of all the enrolled subjects who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab Plus FOLFIRI | Cetuximab Plus FOLFOX | Total
Number analyzed (Participants) | 101 | 188 | 289
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 145 | 215
  >=65 years | 31 | 43 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 69 | 104
  Male | 66 | 119 | 185

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Best Overall Confirmed Response Rate (BORR)
Description: Response rate was defined as the percentage of subjects with BORR (confirmed complete response [CR] or partial response [PR]) according to Response Evaluation Criteria in Solid Tumors (RECIST version 1.0) criteria. As per RECIST v 1.0 criteria for target lesions and assessed by magnetic resonance imaging (MRI): CR = disappearance of all target lesions; PR = at least 30 percent (%) decrease in the sum of the longest diameter of target lesions. Response rate will be assessed every 8 weeks.
Time Frame: From the start of the trial until disease progression, death or last tumor assessment, reported between day of first subject recruited until data cut-off date (31 May 2012)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of subjects
Arm/Group | Cetuximab Plus FOLFIRI | Cetuximab Plus FOLFOX
Number analyzed (Participants) | 101 | 188
Percentage of subjects | 54.5 | 61.2
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs Cetuximab Plus FOLFOX; Test type: Superiority or Other; Odds Ratio (OR) = 1.3176, 95% CI 2-sided [0.8078 to 2.1491]

2. Secondary Outcome: Progression-Free Survival (PFS) Time
Description: PFS time was defined as the time from first administration of study drug until first observation of disease progression or death when death occurs within 90 days of the last tumor assessment or first study drug dose whichever occurred.
Time Frame: From the start of the trial until disease progression, death or last tumor assessment, reported between day of first subject recruited and until data cut-off date (31 March 2014)
Population: The ITT population consisted of all the enrolled subjects who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFIRI | Cetuximab Plus FOLFOX
Number analyzed (Participants) | 101 | 188
months | 11.1 [8.1 to 14.8] | 11.1 [9.0 to 12.7]

3. Secondary Outcome: Overall Survival (OS) Time
Description: OS time was defined as the time from first administration of study drug until date of death, assessed up to 5 years. OS time was censored if the subject was found to be alive on the last date of the assessment.
Time Frame: as for outcome 2
Population: The ITT population consisted of all the enrolled subjects who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFIRI | Cetuximab Plus FOLFOX
Number analyzed (Participants) | 101 | 188
months | 26.6 [21.5 to 33.8] | 27.0 [22.8 to 30.1]

4. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (SAEs), TEAEs Leading to Discontinuation and TEAEs Leading to Death
Description: An Adverse Event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A Serious Adverse Event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: as for outcome 2
Population: Safety population consisted of all the enrolled subjects who received at least one dose of study treatment.
Measure: Number; unit: Subjects
Arm/Group | Cetuximab Plus FOLFIRI | Cetuximab Plus FOLFOX
Number analyzed (Participants) | 101 | 188
Subjects
  TEAEs | 99 | 180
  Treatment Emergent SAEs | 37 | 64
  TEAEs Leading to Death | 5 | 10
  TEAEs Leading to Discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of the trial treatment up to the data cut-off date (31 March 2014)
Description: A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Groups:
- Cetuximab Plus FOLFIRI: Cetuximab was administered intravenously at a dose of 500 milligram per square meter (mg/m^2) biweekly until disease progression, death, or consent withdrawal. Irinotecan was administered intravenously at a dose of 180 mg/m^2 along with folinic acid intravenously at a dose of 400 mg/m^2 (racemic) or 200 mg/m^2 (L-form) and 5-fluorouracil at a dose of 400 mg/m^2 bolus followed by a 46-hour continuous infusion of 2,400 mg/m^2 given biweekly until disease progression, death, or consent withdrawal.
- Cetuximab Plus FOLFOX: Cetuximab was administered intravenously at a dose of 500 milligram per square meter (mg/m^2) biweekly until disease progression, death, or consent withdrawal. Oxaliplatin was administered intravenously at a dose of 100 mg/m^2 along with folinic acid intravenously at a dose of 400 mg/m^2 (racemic) or 200 mg/m^2 (L-form) and 5-fluorouracil at a dose of 400 mg/m^2 bolus followed by a 46-hour continuous infusion of 2,400 mg/m^2 given biweekly until disease progression, death, or consent withdrawal.
Arm/Group | Cetuximab Plus FOLFIRI | Cetuximab Plus FOLFOX
Serious Adverse Events (participants affected / at risk) | 37/101 | 64/188
Other Adverse Events (participants affected / at risk) | 93/101 | 177/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus FOLFIRI (N=101) | Cetuximab Plus FOLFOX (N=188)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 6
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Gastritis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 3 | 0
Intestinal obstruction (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal obstruction (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4
Chest discomfort (General disorders) | 1 | 0
Death (General disorders) | 1 | 2
Disease progression (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 7
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 3
Bacteraemia (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 1
Catheter site infection (Infections and infestations) | 0 | 3
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Mycobacterium abscessus infection (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 0 | 3
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumor perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 0 | 2
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus FOLFIRI (N=101) | Cetuximab Plus FOLFOX (N=188)
Neutropenia (Blood and lymphatic system disorders) | 53 | 100
Leukopenia (Blood and lymphatic system disorders) | 24 | 28
Anaemia (Blood and lymphatic system disorders) | 14 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 44
Cardiac disorders (Cardiac disorders) | 10 | 8
Eye disorders (Eye disorders) | 9 | 20
Nausea (Gastrointestinal disorders) | 61 | 68
Diarrhoea (Gastrointestinal disorders) | 58 | 79
Vomiting (Gastrointestinal disorders) | 37 | 63
Stomatitis (Gastrointestinal disorders) | 31 | 52
Constipation (Gastrointestinal disorders) | 22 | 42
Abdominal pain (Gastrointestinal disorders) | 20 | 14
Mouth ulceration (Gastrointestinal disorders) | 10 | 19
Dyspepsia (Gastrointestinal disorders) | 10 | 10
Abdominal pain upper (Gastrointestinal disorders) | 6 | 12
Abdominal distension (Gastrointestinal disorders) | 6 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 5
Fatigue (General disorders) | 21 | 48
Pyrexia (General disorders) | 17 | 34
Mucosal inflammation (General disorders) | 15 | 54
Asthenia (General disorders) | 7 | 14
Hepatic function abnormal (Hepatobiliary disorders) | 6 | 9
Drug hypersensitivity (Immune system disorders) | 1 | 17
Paronychia (Infections and infestations) | 32 | 48
Upper respiratory tract infection (Infections and infestations) | 11 | 14
Conjunctivitis (Infections and infestations) | 5 | 19
Nasopharyngitis (Infections and infestations) | 1 | 11
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 9 | 15
Weight decreased (Investigations) | 9 | 10
Alanine aminotransferase increased (Investigations) | 6 | 14
Aspartate aminotransferase increased (Investigations) | 3 | 14
Platelet count decreased (Investigations) | 0 | 10
Decreased appetite (Metabolism and nutrition disorders) | 33 | 51
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 29
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 8
Dizziness (Nervous system disorders) | 9 | 23
Headache (Nervous system disorders) | 6 | 14
Dysgeusia (Nervous system disorders) | 6 | 13
Neuropathy peripheral (Nervous system disorders) | 4 | 63
Hypoaesthesia (Nervous system disorders) | 3 | 14
peripheral sensory neuropathy (Nervous system disorders) | 1 | 34
Insomnia (Psychiatric disorders) | 13 | 20
Renal and urinary disorders (Renal and urinary disorders) | 7 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 15
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 17
Rash (Skin and subcutaneous tissue disorders) | 55 | 115
Alopecia (Skin and subcutaneous tissue disorders) | 30 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 29
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 24
Acne (Skin and subcutaneous tissue disorders) | 16 | 22
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 12 | 21
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 | 30
Skin fissures (Skin and subcutaneous tissue disorders) | 11 | 11
Phlebitis (Vascular disorders) | 1 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other